CLINICAL TRIAL: NCT02811627
Title: Predicting Treatment Response to Memantine in Autism Spectrum Disorder Using MR Spectroscopy
Brief Title: Predicting Treatment Response to Memantine in Autism Using Magnetic Resonance Spectroscopy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, David Beversdorf, Assoc. Professor - Medicine: Radiology, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2004983HS
Record Dates: First submitted 2016-06-20; First posted 2016-06-23 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Magnetic Resonance Spectroscopy; Memantine; Treatment prediction biomarker
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Memantine; Magnetic Resonance Imaging

ARMS (1):
- Memantine and Magnetic Resonance Imaging (Experimental): Subjects will be started on memantine post the imaging session.
  Memantine is available commercially as Namenda, Namenda XR and in the liquid form (for subjects who do not wish to take pills). Namenda (pill and the liquid) will be started at 5 mg/day doses to be titrated up 20 mg/day based on response and tolerability, as per the package insert instructions and based upon clinical titration in other clinical trials for a period of 12 weeks. Namenda XR will be started at 7 mg/day to be titrated up to 28mg/day based on response and tolerability, as per package insert instructions and based upon clinical titration in other clinical trials for a period of 12 weeks.
  Interventions: Drug: Memantine; Device: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Memantine — Namenda (pill and the liquid) will be started at 5 mg/day doses to be titrated up 20 mg/day based on response and tolerability, as per the package insert instructions and based upon clinical titration in other clinical trials for a period of 12 weeks. Namenda XR will be started at 7 mg/day to be titrated up to 28mg/day based on response and tolerability, as per package insert instructions and based upon clinical titration in other clinical trials for a period of 12 weeks.
  Other Names: Namenda
Device: Magnetic Resonance Imaging — The subjects will undergo an MRI assessment after baseline behavioral assessment. The session will involve a structural MRI scan, single voxel spectroscopy scans and resting state functional MRI. The subjects will be started on memantine post the imaging session. The imaging will be carried out on a research dedicated 3 Tesla (3T) Siemens Trio Scanner at the University of Missouri Brain Imaging Center by trained personnel.

SUMMARY:
Memantine, an N-methyl-D-aspartate receptor antagonist, has been explored as a possible therapeutic agent that reduces the excitatory (glutamate) - inhibitory (gamma amino-butyric acid, GABA) imbalance in autism pathology and improves social and communication deficits. While some studies have shown positive results, a large clinical trial failed to show benefit possibly because different subsets of autism responded differently to the treatment.

The investigator proposes a pilot, exploratory, clinical follow-on study using proton magnetic resonance spectroscopy (1H-MRS) to determine whether baseline glutamate/GABA levels in certain regions of the brain may help predict treatment response to Memantine in autistic subjects. At study onset, subjects will be assessed on the behavioral scales such as the Aberrant Behavior Checklist and Clinical Global Impressions scale, followed by MRS imaging. Memantine treatment will be started post imaging. Assessment measures will be repeated at week 12 during treatment. Glutamate and GABA levels in brain regions will be correlated to improvements on assessment measures. Expected results include higher glutamate and/or lower GABA levels in the anterior cingulate cortex at baseline in responders to memantine. If the hypotheses are confirmed, it will provide evidence of a relevant neural biomarker to predict treatment response to memantine with important implications for clinical care including improving individualization of treatments.

DETAILED DESCRIPTION:
Background and Rationale

Autism Spectrum Disorder (ASD) is a behaviorally defined complex neurodevelopmental disorder characterized by early childhood onset of marked deficiencies in social and communication skills and presence of restrictive, repetitive behaviors. Its phenotypic heterogeneity makes studying ASD and its treatment a challenging task. Currently, only two FDA approved drugs, risperidone and aripiprazole, are available to treat ASD that manage irritability associated with the disorder. None have shown conclusive benefit for core features of social and communication deficits.

Research indicates that a disrupted balance between excitation (glutamate) and inhibition (gamma amino-butyric acid, GABA) is likely to be one of the underlying mechanisms of ASD. This hypothesis is supported by a number of magnetic resonance spectroscopy studies that report an excess of glutamatergic excitation and/or a reduction in GABAergic inhibition observed in different brain regions including the limbic system and the anterior cingulate cortex. Similar findings have also been reported in post mortem studies of the ASD brain.Thus, it is expected that drugs targeting this imbalance could be beneficial. For example, the GABAB agonist, arbaclofen, was tested in ASD for this reason and showed promising results but a large trial failed to show improvement on the primary endpoints of lethargy and social withdrawal.

Memantine, a moderate affinity N-methyl-D-aspartate (NMDA) receptor antagonist, is known to improve communication in patients with Alzheimer's disease and is an FDA approved treatment for that disease. Examination of the efficacy of memantine in treating ASD has also been driven by the excitatory (glutamate) - inhibitory (gamma amino-butyric acid, GABA) imbalance hypothesis of ASD pathology. Memantine binds to the glutamatergic NMDA receptors and attenuates glutamatergic excitation. This reduction in excessive glutamatergic activation is thought to decrease the "noise" in the neural network system and facilitate learning and memory. A few small studies have shown effectiveness for memantine in the treatment of social and communication aspects of ASD spectrum disorder (ASD) as well. However, one large clinical trial using memantine in ASD reported a failure to respond. These discrepancies in results could possibly be due to the heterogeneity in the excitatory-inhibitory imbalance between ASD patients thereby causing a variation in response. In such a scenario, having a biomarker to predict an individual's treatment response would be invaluable.

MR Spectroscopy is a non-invasive tool used to examine the biochemical profile of brain tissue associated with different psychiatric and neurological conditions including ASD. Specifically, 1H-MRS studies in ASD demonstrated the excitatory-inhibitory imbalance in various cortical and subcortical regions of the brain, a finding also reported in post mortem brain tissue studies. The use of this technique to determine if Glutamate/GABA concentrations in certain regions of the brain can predict response to treatment with memantine would be an innovative breakthrough in providing more effective individualized treatment for patients since very little research has been done to explore this possibility.

A similar approach has been adopted in a recent ongoing study that uses proton MR spectroscopy to map changes in glutamate and GABA following use of riluzole in ASD. Riluzole is a drug commonly used in amyotrophic lateral sclerosis (ALS) and is a glutamate antagonist that works by blocking presynaptic glutamate release and noncompetitive inhibition of NMDA receptors. However, riluzole is not clinically used in the treatment of ASD. To our knowledge, only one study so far (apart from the ongoing study mentioned) has examined the effects of riluzole in ASD, but as an adjunct to risperidone. The primary outcomes of the Ghaleiha et al. study were irritability and repetitive motor behaviors and not core social and communication deficits as in the present proposal. The purpose of riluzole in this MR spectroscopy study is a proof of principle for its effects on spectroscopy based on its glutamate antagonistic effects. By contrast, memantine, which will be studied in the present proposal, has some documented evidence from small studies of being beneficial in treating social and communication deficits associated with ASD in clinical settings, despite the failure of the larger trial.

The investigator's lab has previously utilized MR spectroscopy techniques to map these different compounds in a group of 14 subjects with ASD and identify glutamate and GABA alterations in the cerebellum, discovering a relationship to cerebrocerebellar connectivity and behavioral outcomes in individuals with ASD.

Specific Aims:

Specific Aim 1: The investigator proposes a pilot, exploratory, clinical follow-on study using proton magnetic resonance spectroscopy (1H-MRS) to examine whether the following measures can be used to predict treatment response to memantine in ASD:

1. Glx and/or GABA and the Glx/GABA ratio in the anterior cingulate cortex,
2. Glx levels in the dorsolateral prefrontal cortex and the cerebellum
3. Markers of neuronal integrity, N-acetyl aspartate (NAA), myo-inositol, choline and creatine/phosphocreatine levels in the anterior cingulate, dorsolateral prefrontal cortex and cerebellum

Specific Aim 2: To examine whether resting state functional connectivity between the dorsolateral prefrontal cortex, anterior cingulate and the cerebellum, holds predictive value for treatment response to memantine in ASD.

The anterior cingulate cortex, dorsolateral prefrontal cortex and the cerebellum have been have been chosen as regions of interest (ROIs) due to known atypical glutamate and GABAergic profiles in these regions associated with ASD. The approach of limiting to selected ROIs has been adopted in order to ensure patient comfort during the imaging process by reducing the time spent in the scanner. Since altered levels for markers of neuronal integrity, such as NAA, choline, creatine/phosphocreatine and myoinositol have also been reported in ASD, we will be mapping these biochemicals as well in order to explore their effect on treatment response. Resting state functional connectivity will also be analyzed for possible association with treatment outcome prediction since as mentioned before, a previous study from the investigator's has shown a link between alterations in resting state cerebrocerebellar connectivity, excitatory-inhibitory ratio in the cerebellum and behavioral outcome in ASD using MR spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants will be asked to take part in this study because he/she:

  1. has autism spectrum disorder
  2. is starting memantine off label for managing their autism symptoms
  3. is deemed safe to enter the MR environment using the attached screening form, and
  4. is capable of lying still for approximately 1.5 hour.

Exclusion Criteria:

* Subjects would be excluded if:

  1. they have certain types of metallic implants, risk of exposure to metallic foreign bodies, pacemakers, magnetically sensitive implants that cannot be removed or are not securely attached,
  2. pregnancy
  3. claustrophobia
  4. memantine intolerance
  5. known hypersensitivity to memantine hydrochloride or
  6. inability to lie still for approximately 90 minutes.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impressions - Improvement | 12 weeks post start of memantine treatment
  Clinician rated 7 item scale looking at improvements in specific aspects and overall level of autism

SECONDARY OUTCOMES:
Social Responsiveness Scale (SRS) | Baseline (before start of memantine treatment) and at 12 weeks post start of memantine treatment
  Assessment of baseline social deficits before treatment onset and improvement in social functioning 12 weeks after starting memantine treatment. The Social Responsiveness Scale (SRS) is a 65 item questionnaire rated on a 4 point Likert scale to evaluate social impairments in autism. Higher scores on the SRS indicate severe impairments in social skills while lower scores indicate mild to moderate impairment in social skills. Total raw score pre and post treatment will be compared.
General Social Outcomes Measure (GSOM) | Baseline (before start of memantine treatment) and at 12 weeks post start of memantine treatment
  The General Social Outcomes Measure assesses individuals with autism on five sub scales including Conversational Reciprocity, Social Problem solving, Affect Demonstration and Emotional Perspective Taking. Assessment of baseline social deficits before treatment onset and improvement in social functioning 12 weeks after starting memantine treatment. Lower scores indicate more severe impairment of social deficits while higher scores indicate improvements in social functioning. Scores on individual sub scales pre and post treatment will be compared.
Aberrant Behavior Checklist (ABC) | Baseline (before start of memantine treatment) and at 12 weeks post start of memantine treatment
  Assessment of baseline and post-treatment levels of irritability, lethargy/social withdrawal, stereotypic behavior, hyperactivity or noncompliance and inappropriate speech. Higher scores indicate greater impairments.
Test of Language Competence | Baseline (before start of memantine treatment) and at 12 weeks post start of memantine treatment
  Assesses language comprehension and verbal skills. Includes multiple sub tests such as Ambiguous Sentences, Figurative Speech and Recreating Oral Expressions. Higher scores indicate low levels of impairment in the domain. Scores on the individual sub scales will be compared pre and post treatment to assess improvements.

CONTACTS AND LOCATIONS:
Overall Officials: David Q Beversdorf, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT02811627/Prot_SAP_000.pdf